CLINICAL TRIAL: NCT07208838
Title: Validation of DDIVAT Digital Optotypes for Distance Visual Acuity Testing Among the Bulgarian Population
Status: Enrolling by invitation | Type: Observational
Sponsor: Plovdiv Medical University (Other)
Collaborators: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Vasil Marinov, MD, PhD, Plovdiv Medical University
Other Study IDs: PlovdivMUDDIVAT
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-04

CONDITIONS: Vision Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: 75 males and 75 females over 18 years of age
  Interventions: Diagnostic Test: To test visual acuity in 150 Bulgarian patients over 18 years of age using Snellens visual acuity chart and DDIVAT optotypes

INTERVENTIONS:
Diagnostic Test: To test visual acuity in 150 Bulgarian patients over 18 years of age using Snellens visual acuity chart and DDIVAT optotypes — The study compares newly developed visual acuity test (DDIVAT) with standart method for visual acuity testing used worldwide

SUMMARY:
To compare distance visual acuity in Bulgarian patients over 18 years of age using two different methods - the Snellen method and the DIDIVAT digital online optotypes. For the purpose of this study, it is planned to examine native visual acuity (with and without prescribed optical correction), without additional mydriasis in both ways, of 150 Bulgarian patients (75 women and 75 men) over 18 years of age, hospitalized in a university eye clinic at St. George University Hospital and healthy volunteers willing to participate in the study. The statistical analysis that will be performed will aim to compare whether the two methods for determining distance visual acuity are identical in results, as well as to validate the application for the Bulgarian population.The study is expected to prove that the distance visual acuity of patients examined by both methods is identical.

ELIGIBILITY:
Inclusion Criteria:

* Bulgarian speaking patients (75 women and 75 men) over 18 years of age, hospitalized in a university eye clinic at St. George University Hospital and healthy volunteers willing to participate in the study.

Exclusion Criteria:

* Patients of less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bulgarian speaking patients (75 women and 75 men) over 18 years of age, hospitalized in a university eye clinic at St. George University Hospital and healthy volunteers willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The study is expected to prove that the distance visual acuity of patients examined by both methods is identical. | 12 monts

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Plovdiv, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bakirtzis M, Michaleakou E, Martidou ME, Lahana E, Kostagiolas P, Niakas D, Labiris G. Visual Acuity Screening of Refugees and Immigrants with a Web-Based Digital Test: A Pilot Study. Acta Medica (Hradec Kralove). 2024;67(3):79-86. doi: 10.14712/18059694.2025.2. PMID 39963735
- [Background] Labiris G, Panagiotopoulou EK, Duzha E, Tzinava M, Perente A, Konstantinidis A, Delibasis K. Development and Validation of a Web-Based Reading Test for Normal and Low Vision Patients. Clin Ophthalmol. 2021 Sep 22;15:3915-3929. doi: 10.2147/OPTH.S314943. eCollection 2021. PMID 34588763
- [Background] Labiris G, Panagiotopoulou EK, Chatzimichael E, Tzinava M, Mataftsi A, Delibasis K. Introduction of a digital near-vision reading test for normal and low vision adults: development and validation. Eye Vis (Lond). 2020 Oct 22;7:51. doi: 10.1186/s40662-020-00216-0. eCollection 2020. PMID 33102611
- [Background] Labiris G, Panagiotopoulou EK, Delibasis K, Duzha E, Bakirtzis M, Panagis C, Boboridis K, Mokka A, Balidis M, Damtsi C, Ntonti P. Validation of a web-based distance visual acuity test. J Cataract Refract Surg. 2023 Jul 1;49(7):666-671. doi: 10.1097/j.jcrs.0000000000001176. PMID 36853857